CLINICAL TRIAL: NCT04329832
Title: Hydroxychloroquine vs. Azithromycin for Hospitalized Patients With Suspected or Confirmed COVID-19 (HAHPS): A Prospective Pragmatic Trial
Brief Title: Hydroxychloroquine vs. Azithromycin for Hospitalized Patients With Suspected or Confirmed COVID-19
Acronym: HAHPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Samuel Brown, Director, Critical Care Research, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1051355
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Hydroxychloroquine; Azithromycin
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental)
  Interventions: Drug: Hydroxychloroquine
- Azithromycin (Active Comparator)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Hydroxychloroquine — Patients in the hydroxychloroquine arm will receive hydroxychloroquine 400 mg by mouth twice daily for 1 day, then 200 mg by mouth twice daily for 4 days (dose reductions for weight < 45 kg or GFR (glomerular filtration rate)<50ml/min). For patients < 45kg, doses will be halved. For patients with GFR<50ml/min, the final dose of hydroxychloroquine will not be administered. If the patient has already received hydroxychloroquine prior to randomization (no more than 2 days), the prior doses will count toward the 5-day total.
  Arms: Hydroxychloroquine
Drug: Azithromycin — Patients in the azithromycin arm will receive azithromycin 500 mg on day 1 plus 250 mg daily on days 2-5 (may be administered intravenously per clinician preference). If the patient has already received azithromycin prior to randomization (no more than 2 days), the prior doses will count toward the 5-day total.
  Arms: Azithromycin

SUMMARY:
This study will compare two drugs (hydroxychloroquine and azithromycin) to see if hydroxychloroquine is better than azithromycin in treating hospitalized patients with suspected or confirmed COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years)
* Confirmed OR suspected COVID-19,

  * Confirmed: Positive assay for COVID-19 within the last 10 days
  * Suspected: Pending assay for COVID-19 WITH high clinical suspicion
* Scheduled for admission or already admitted to an inpatient bed

Exclusion Criteria:

* Allergy to hydroxychloroquine or azithromycin
* History of bone marrow transplant
* Known G6PD deficiency
* Chronic hemodialysis or Glomerular Filtration Rate < 20ml/min
* Psoriasis
* Porphyria
* Concomitant use of digitalis, flecainide, amiodarone, procainamide, propafenone, cimetidine, dofetilide, phenobarbital, phenytoin, or sotalol
* Known history of long QT syndrome
* Current known QTc>500 msec
* Pregnant or nursing
* Prisoner
* Weight < 35kg
* Seizure disorder
* Severe liver disease
* Outpatient use of hydroxychloroquine for treatment of a disease other than COVID-19 OR has received more than 2 days of hydroxychloroquine or azithromycin for suspected or confirmed COVID-19
* Patient has recovered from COVID-19 and/or is being discharged from the hospital on day of enrollment.
* Treating physician refuses to allow patient participation in the study
* Unable to obtain informed consent
* Prior enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel M Brown, MD MS, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
In order to protect patient privacy and comply with relevant regulations, identified data are unavailable. Requests for deidentified data from qualified researchers with appropriate ethics board approvals and relevant data use agreements will be processed by the Intermountain Office of Research, officeofresearch@imail.org.

REFERENCES:
- [Background] WHO, 2020. WHO R&D Blueprint, novel Coronavirus, COVID-19 Therapeutic Trial Synopsis. https://www.who.int/publications/i/item/covid-19-therapeutic-trial-synopsis
- [Derived] Koric A, Chang CP, Mark B, Rowe K, Snyder J, Dodson M, Deshmukh VG, Newman MG, Fraser AM, Smith KR, Date AP, Gren LH, Porucznik CA, Haaland BA, Henry NL, Hashibe M. Cardiovascular disease risk in long-term breast cancer survivors: A population-based cohort study. Cancer. 2022 Jul 15;128(14):2826-2835. doi: 10.1002/cncr.34224. Epub 2022 May 13. PMID 35561317
- [Derived] Brown SM, Peltan I, Kumar N, Leither L, Webb BJ, Starr N, Grissom CK, Buckel WR, Srivastava R, Butler AM, Groat D, Haaland B, Ying J, Harris E, Johnson S, Paine R 3rd, Greene T. Hydroxychloroquine versus Azithromycin for Hospitalized Patients with COVID-19. Results of a Randomized, Active Comparator Trial. Ann Am Thorac Soc. 2021 Apr;18(4):590-597. doi: 10.1513/AnnalsATS.202008-940OC. PMID 33166179
- [Derived] Brown SM, Peltan ID, Webb B, Kumar N, Starr N, Grissom C, Buckel WR, Srivastava R, Harris ES, Leither LM, Johnson SA, Paine R 3rd, Greene T. Hydroxychloroquine versus Azithromycin for Hospitalized Patients with Suspected or Confirmed COVID-19 (HAHPS). Protocol for a Pragmatic, Open-Label, Active Comparator Trial. Ann Am Thorac Soc. 2020 Aug;17(8):1008-1015. doi: 10.1513/AnnalsATS.202004-309SD. PMID 32425051
- See also: Source for WHO COVID Ordinal Outcomes Scale — https://www.who.int/publications/i/item/covid-19-therapeutic-trial-synopsis

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxychloroquine | Azithromycin
Started | 42 | 43
Completed | 42 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Azithromycin | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [42 to 60] | 58 [43 to 68] | 55 [42 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 23 | 29 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 32
  Not Hispanic or Latino | 25 | 28 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 8
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 6 | 4 | 10
  Black or African American | 1 | 0 | 1
  White | 26 | 28 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 42 | 43 | 85
Comorbidities [Median (Inter-Quartile Range); unit: Scores on a scale] — The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes found in administrative data, such as hospital abstracts data. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of 0 indicates no comorbidities were found. The higher the score (max 24) the more likely the predicted outcome will result in mortality or higher resource use.
  Scores on a scale | 1 [0 to 2] | 0 [0 to 2] | 1 [0 to 2]

OUTCOME MEASURES:

1. Primary Outcome: COVID Ordinal Outcomes Scale at 14 Days
Description: Improvement of clinical condition of the patient defined by the COVID-19 WHO ordinal Outcomes score. This scale reflects a range from uninfected to dead, where 0 is "no clinical or virological evidence of infection", 1 is "no limitation of activities", 2 is "limitation of activities", 3 is "hospitalized, no oxygen therapy", 4 is "oxygen by mask or nasal prongs", 5 is "non-invasive ventilation or high-flow oxygen", 6 is "intubation and mechanical ventilation", 7 is "ventilation + additional organ support - pressors, RRT (renal replacement therapy), ECMO (extracorporeal membrane oxygenation)", and 8 is "death".
Time Frame: Assessed once on day 14 after enrollment (enrollment is day 0)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Day 14 WHO COVID Score: Hydroxychloroquine: The median WHO COVID Score at Day 14 for patients in the hydroxychloroquine arm
- Day 14 WHO COVID Score: Azithromycin: The median WHO COVID Score at Day 14 for patients in the azithromycin arm
Arm/Group | Day 14 WHO COVID Score: Hydroxychloroquine | Day 14 WHO COVID Score: Azithromycin
Number analyzed (Participants) | 42 | 43
score on a scale | 2.0 [2.0 to 3.75] | 2.0 [1.5 to 3.0]

2. Secondary Outcome: Hospital-free Days at 28 Days
Description: Calculated as number of days patient not in hospital
Time Frame: Admission (day 1) to 28 days after admission (day 28)
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Hydroxychloroquine: The median number of hospital-free days for hydroxychloroquine (Interquartile range)
- Azithromycin: The median number of hospital-free days for azithromycin (Interquartile range)
Arm/Group | Hydroxychloroquine | Azithromycin
Number analyzed (Participants) | 42 | 43
Days | 18.5 [7.25 to 24.75] | 21 [7.5 to 24]

3. Secondary Outcome: Ventilator-free Days at 28 Days (Number of Days Patient Not on a Ventilator)
Description: Calculated as number of days that patient is not on a ventilator up to day 28 days after admission
Time Frame: Admission (day 1) to 28 days after admission (day 28)
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Ventilator-Free Days at Day 28 for Hydroxychloroquine Arm: Number of days that the patient is not on a ventilator up to 28 days following admission for patients in the Hydroxychloroquine Arm
- Ventilator-Free Days at Day 28 for Azithromycin Arm: Number of days that the patient is not on a ventilator up to 28 days following admission for patients in the Azithromycin Arm
Arm/Group | Ventilator-Free Days at Day 28 for Hydroxychloroquine Arm | Ventilator-Free Days at Day 28 for Azithromycin Arm
Number analyzed (Participants) | 42 | 43
days | 18 [10.75 to 18] | 18 [12 to 18]

4. Secondary Outcome: ICU-free Days at 28 Days
Description: Calculated as number of days patient not in an ICU
Time Frame: Admission (day 1) to 28 days after admission (day 28)
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Hydroxychloroquine: The median ICU-free days for hydroxychloroquine (Interquartile Range)
- Azithromycin: The median ICU-free days for azithromycin (Interquartile Range)
Arm/Group | Hydroxychloroquine | Azithromycin
Number analyzed (Participants) | 42 | 43
Days | 18 [8 to 22] | 19 [8.5 to 22]

5. Secondary Outcome: Time to a 1-point Decrease in the WHO Ordinal Recovery Score
Description: Time to 1-point decrease in the WHO ordinal recovery score is defined as the number of days until the ordinal outcome score drops by 1 relative to baseline on the 8-point WHO COVID Ordinal Outcomes scale, which reflects a range from uninfected to dead, where 0 is "no clinical or virological evidence of infection", 1 is "no limitation of activities", 2 is "limitation of activities", 3 is "hospitalized, no oxygen therapy", 4 is "oxygen by mask or nasal prongs", 5 is "non-invasive ventilation or high-flow oxygen", 6 is "intubation and mechanical ventilation", 7 is "ventilation + additional organ support - pressors, RRT (renal replacement therapy), ECMO (extracorporeal membrane oxygenation)", and 8 is "death".
Time Frame: Admission (day 1) to 14 days after admission (day 14)
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Days to a 1-point Decrease in WHO COVID Scale in Hydroxychloroquine Arm: Time (in days) until the ordinal outcome score drops by 1 relative to baseline on the 8-point WHO COVID Ordinal Outcomes scale for patients in the Hydroxychloroquine Arm.
- Days to a 1-point Decrease in WHO COVID Scale in Azithromycin Arm: Time (in days) until the ordinal outcome score drops by 1 relative to baseline on the 8-point WHO COVID Ordinal Outcomes scale for patients in the Azithromycin Arm.
Arm/Group | Days to a 1-point Decrease in WHO COVID Scale in Hydroxychloroquine Arm | Days to a 1-point Decrease in WHO COVID Scale in Azithromycin Arm
Number analyzed (Participants) | 42 | 43
Days | 7 [3 to 13] | 6 [2.5 to 10]

ADVERSE EVENTS:
Time Frame: Hospital discharge of the specific subject. Median length of stay for patients in both arms is 7.8 days. Upper bound of IQR for Hydroxychloroquine arm is 15.55 days and upper bound of IQR for Azithromycin arm is 20.85 days.
Arm/Group | Hydroxychloroquine | Azithromycin
All-Cause Mortality (participants affected / at risk) | 6/42 | 1/43
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 3/42 | 2/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=42) | Azithromycin (N=43)
QT Prolongation (Cardiac disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT04329832/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT04329832/SAP_001.pdf